CLINICAL TRIAL: NCT06386172
Title: An Electronic Triggering Decision-support System to Improve Detection, Management and Nephrologist Referral of Patients With Chronic Kidney Disease in Primary Care: A Pragmatic Cluster Randomized Controlled Trial
Brief Title: Electronic Decision-support System to Improve Detection and Care of Patients With Chronic Kidney Disease in Stockholm
Acronym: ALMA-CKD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Danderyd Hospital (Other); Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Juan Jesus Carrero, Professor of Cardiorenal Epidemiology, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023-03537-01; FoUI-986028 (Other Grant/Funding Number: ALF Medicin, Region Stockholm)
Record Dates: First submitted 2024-01-26; First posted 2024-04-26 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Chronic Kidney Diseases
Keywords: Chronic Kidney Disease; Clinical Decision Support system; Pragmatic cluster-Randomized controlled trial; SCREAM; Guidelines, processes of care
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: The primary healthcare network system of the region of Stockholm coordinates 66 public primary healthcare centers. Collectively, these centers offer care to an estimated population of 780.000. Since November 2022, a new platform for CDS (clinical decision support) triggers called ALMA has been implemented in these centers. ALMA is connected to patient records and uses CDS triggers to identify medical problems, issue alerts and propose solutions.
  Using the ALMA platform, this project has the following objectives:
  Objective 1: to develop a CDS trigger connected with the electronic healthcare records specific to the processes of screening, diagnosis, and nephrologist referral of patients with CKD, including individualized CKD management optimization, in primary care.
  Objective 2: to evaluate the effectiveness of this CDS trigger (versus current basic advice) through a 2-arm pragmatic cluster RCT.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Centers which have been randomized to recieve the intervention with CKD clinical decision support triggers will be administered via ALMA
  Interventions: Other: Clinical decision support trigger
- Care as usual (No Intervention): Centers which have been randomized to no intervention and receive only prior/general clinical decision support triggers currently available in the ALMA platform. They do not receive the specific clinical decision support triggers for CKD.

INTERVENTIONS:
Other: Clinical decision support trigger — Investigation of CDS-triggers effect on primary care physicians detection and management of chronic kidney disease
  Arms: Intervention

SUMMARY:
One in 10 adults in Region Stockholm have chronic kidney disease (CKD), which dramatically increases healthcare costs and the risk of medication errors or adverse health outcomes, including cardiovascular disease and death. Identification and early management of these patients is done in primary care settings. However, most adults with CKD in our region are under detected, undiagnosed and undertreated, with low rates of referral to nephrology-specialist care.

This is a pragmatic cluster randomized controlled trial (RCT) involving 66 primary healthcare centers in Region Stockholm, and testing the effect of an electronic clinical decision support (CDS) triggering system to assist general practitioners through the guideline-recommended processes of CKD care.

The centers, providing healthcare to approximately 780.000 citizens, will be randomized 50:50 to this CDS trigger (vs basic advice) for 18 months. Study outcomes will consider the improvement in the indicators of CKD care.

As a pragmatic trial there is no active recruitment or active data collection. The trial is embedded into the ongoing Stockholm CREAtinine Measurements (SCREAM) project, a database collection of healthcare use for the complete population of Stockholm. Using this real-world healthcare data collection, the investigators will be able to measure with precision the impact of our CDS trigger and its potential to improve clinical care.

DETAILED DESCRIPTION:
A large proportion of persons in our region suffer from CKD and are not adequately identified and cared for.

The hypothesis tested in this trial is that providing a structured framework of advice in the form of an electronic clinical decision support (CDS) triggering system to general practitioners has the potential to improve the identification, recognition and care of persons with CKD.

About 10% of adults in Stockholm suffer from CKD, a condition characterized by reduced kidney function or signs of kidney damage that are sustained over time. CKD is disproportionally present in older adults (in 18% of persons aged 66-74, and 41% of persons aged >75 years) and in those with non-communicable diseases like hypertension (in 29% of patients), diabetes (26%) and cardiovascular disease (37%).

CKD can be identified and diagnosed with two simple and inexpensive laboratory analyses:

* serum/plasma creatinine, which serves to estimate glomerular filtration rate (eGFR) as a marker of kidney function,
* and albumin in urine (albuminuria), which serves as a marker of kidney damage.

Despite the low cost and widespread availability of these tests, they are not measured or interpreted to a desirable degree in primary health care. This leads to a high degree of under-detection and under-recognition of CKD. In Stockholm, only 9% of people with laboratory-detected CKD carried a clinical diagnosis or visited a nephrologist.

Patients with CKD have increased risks of all-cause mortality, cardiovascular mortality and morbidity, and kidney failure requiring dialysis or transplantation. They are also prone to suffer from medication errors, given that the loss of kidney function requires careful consideration of drug dosages and represents a contraindication for many common therapies. The management of CKD is costly: dialysis and transplantation alone, which affects to only 1-2% of the total population with CKD, typically represents 2-3% of the total healthcare expenditure of developed countries.

Many patients with CKD are at low risk of progression to kidney failure and are ideally managed in primary care settings. This is the current model of decentralized CKD care of most health systems including Region Stockholm. Regional, national and international guidelines provide clear recommendations regarding the screening, identification, management of patients with CKD in primary care as well as criteria for referral to nephrologist care. The goal of these recommendations is to improve detection and recognition, as well as to reduce the risk of adverse consequences of kidney failure and cardiovascular disease.

Despite the presence of clear guidelines, international reports suggest that most adults with CKD remain under detected, undiagnosed, improperly risk stratified, and undertreated. Even when laboratory data is present to substantiate a CKD diagnosis, clinicians often do not recognize or diagnose it, and, as a result, medication errors can occur. Another missed opportunity of poor identification and recognition of CKD is that patients with advanced CKD often are not referred to nephrology early enough to have meaningful discussions about preparation for kidney replacement therapy.

Barriers that hinder effective CKD identification and care in primary care settings include lack of awareness and/or understanding of guidelines for risk stratification and management of CKD, confusion regarding appropriate referral criteria and timing, lack of confidence in managing CKD and limited communication channels with specialists in nephrology. Additionally, general practitioners may have limited time to manage complex visit agendas. Programs that facilitate the processes of CKD identification and management as well as enhanced cooperation between general and specialist care have thus the potential to improve these identified care gaps.

Widespread use of electronic health records offers new opportunities to identify and address such care gaps, by implementation of electronic clinical decision support (CDS) systems. CDS systems are designed to aid clinician decision making during the process of care. When well designed and effectively used, they can be powerful tools for improving the quality of patient care and preventing errors and omissions.

CDS triggers, that is, CDS systems that automatically activate upon a "trigger" (e.g. when the patient journal is opened or a laboratory test is ordered), have advantages compared with CDS systems that require active engagement of the clinician (i.e. having to access a specific website or platform to consult advice). CDS triggers can facilitate actions and promote proactive preventive care, such as opportunistic disease screening; they can also serve as reminders to staff and clinicians to take action to improve care delivery to a patient, alerting them while they're working in the electronic healthcare records, and linking them to the appropriate place to take the preferred action.

Since November 2022, a new platform for CDS triggers called ALMA has been implemented in the 66 public primary healthcare centers of Region Stockholm. ALMA is connected to patient records and uses CDS triggers to identify medical problems, issue alerts and propose solutions. At present, ALMA provides basic advice for the management of CKD, which consists of the recommendation to "measure albuminuria once annually in patients with diabetes". This trial will use the already-established ALMA platform to conduct a pragmatic RCT with the goals above mentioned.

ELIGIBILITY:
Inclusion criteria:

People with conditions for which clinical guidelines recommend annual screening for kidney disease:

* Diabetes
* Hypertension
* People with a chronic kidney disease diagnosis.
* People with a rapidly declining eGFR (loss of 15% in the last 3 months or > 5 ml/min/1.73m2 per year).
* People with albuminuria (>3 mg/mmol)

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2023-09-09 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Number of participants screened for creatinine and albuminuria | Through study completion, an average of 18 months
  The number of eligible persons (i.e with an indication for screening) screened for creatinine and albuminuria once annually. Patients eligible for screening are, according to current guidelines those with hypertension, diabetes or history of cardiovascular disease.
Number of screened participants with retesting for creatinine and albuminuria | Through study completion, an average of 18 months
  The re-testing of these labs within 3-6 months among people with abnormal eGFR (<60 ml/min/1.73 m2) or albuminuria (>30 mg/g) at screening.

SECONDARY OUTCOMES:
Number of participants with laboratory-determined CKD receiving a clinical diagnosis | Through study completion, an average of 18 months
  Among those fulfilling criteria of outcome 2 (i.e. sustained signs of CKD over time), proportion of clinical diagnoses issued
Number of participants receiving CKD-modifying agents | Through study completion, an average of 18 months
  Among people fulfilling criteria 2, proportion of initiation of CKD-modifying agents
Number of participants referred to nephrologist care | Through study completion, an average of 18 months
  Among those fulfilling National Criteria for referral.

CONTACTS AND LOCATIONS:
Overall Officials: Juan J Carrero, Prof, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No
Not allowed by hospital, institutional and GDPR regulations

REFERENCES:
- [Derived] Andersson-Emad J, Thunholm A, Nash S, Evans M, Lind Af Hageby S, Arnlov J, Hilderman M, Forseth M, Sjolander A, Jacobson SH, Carrero JJ. Study protocol of the ALMA-CKD trial; an electronic triggering decision-support system to improve the detection, recognition, and management of patients with chronic kidney disease in primary care. BMC Nephrol. 2024 Nov 13;25(1):408. doi: 10.1186/s12882-024-03852-z. PMID 39538192

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-11-20): https://cdn.clinicaltrials.gov/large-docs/72/NCT06386172/SAP_001.pdf